CLINICAL TRIAL: NCT03559530
Title: Acinetobacter Baumannii-related Osteomyelitis: Clinical and Epidemiological Characterization
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Priscila Rosalba Domingos de Oliveira, Investigator, University of Sao Paulo
Other Study IDs: 14186
Record Dates: First submitted 2018-05-04; First posted 2018-06-18 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Osteomyelitis
Keywords: osteomyelitis; Acinetobacter baumannii; Anti-Infective Agents
MeSH Terms: conditions — Osteomyelitis | interventions — Anti-Infective Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with microbiologically proven A. baumannii-related osteomyelitis
  Interventions: Drug: Antimicrobial

INTERVENTIONS:
Drug: Antimicrobial — Antimicrobial therapy according to A. baumannii susceptibility profile

SUMMARY:
Acinetobacter baumannii is an opportunist pathogen that has become increasingly important over recent years as a cause of nosocomial infections. Ventilator-associated pneumonia, central line-associated bloodstream infection and bone and soft tissue infections secondary to open fractures are among the conditions most associated with this agent .

Attention is drawn not only to the increasing incidence of this agent over the last few years but also to the rapid worsening of its susceptibility to antimicrobial agents, including carbapenems. Few therapeutic options are available for treating pan-resistant strains: colistin and tigecycline has been used, but resistance to these options frequently emerges in clinical practice. Taking into account the fact that fewer new antimicrobial agents are being validated and introduced into clinical practice, the growing prevalence of isolates with these high levels of resistance is becoming a matter of increasing concern.

Certain risk factors have also been correlated with infection related to A. baumannii. The most important are prolonged hospitalization in intensive care units and use of invasive devices. Another important risk factor is severe trauma: A. baumannii is associated with invasive infections, including osteomyelitis following open fracture reduction. Studies that included military personnel and civilians involved in the recent conflicts in Iraq and Afghanistan have shown high prevalence of A. baumannii as causative agent in cases of osteomyelitis secondary to traumatic injuries. Also, in Brazil, a retrospective study that analyzed 101 cases of osteomyelitis due to Gram-negative bacilli showed that A. baumannii was the second most prevalent agent and that it had a high degree of antimicrobial resistance, particularly to carbapenems.

The objectives of this retrospective study are: 1. clinically and epidemiologically characterize 241 patients with osteomyelitis related to A. baumannii who were admitted at the Institute of Orthopedics and Traumatology, Hospital das Clínicas, University of São Paulo; 2. to describe the antimicrobial susceptibility profile of A. baumannii strains isolated; 3. to evaluate the patients' outcomes (remission, recurrence, limb amputation or death) according to the antimicrobial treatment used, including tigecycline; 4. to compare efficacy and safety profiles of tigecycline, colistin and ampicillin-sulbactan among patients with carbapenem-resistant A. baumannii related osteomyelitis.

DETAILED DESCRIPTION:
INTRODUCTION Acinetobacter baumannii is an opportunist pathogen that has become increasingly important over recent years as a cause of nosocomial infections (1,2). Ventilator-associated pneumonia, central line-associated bloodstream infection and bone and soft tissue infection secondary to open fractures are among the conditions most associated with this agent.

Attention is drawn not only to the increasing incidence of this agent over the last few years but also to the rapid worsening of its susceptibility to antimicrobial agents, including carbapenems. Among the striking characteristics of this species is its high capacity to develop antimicrobial resistance. The most important types of resistance are, firstly, intrinsic resistance related to the association between diminished permeability of the external membrane and constitutive expression of efflux pumps; and secondly, acquisition of genetic elements, which might be resistance genes or insertion elements that, in association with the chromosomal genes of this bacterium, can trigger expression of resistance and great ability to survive in the environment, which is commonly related to production of biofilm (7). All these characteristics have been correlated with emergence of multiresistant and pan-resistant strains of A. baumannii. Few therapeutic options are available for treating pan-resistant strains: colistin and tigecycline has been used, but resistance to these options frequently emerges in clinical practice. Taking into account the fact that fewer new antimicrobial agents are being validated and introduced into clinical practice, the growing prevalence of isolates with these high levels of resistance is becoming a matter of increasing concern. The formerly abundant flow of provision of new antibiotics of ever-broader spectrum has been shown to be a non-renewable resource.

Certain risk factors have also been correlated with occurrence of A. baumannii. The most important are prolonged hospitalization in intensive care units and use of invasive devices .Another important risk factor is severe trauma: A. baumannii is associated with invasive infections, including osteomyelitis following open fracture reduction. Studies that included military personnel and civilians involved in the recent conflicts in Iraq and Afghanistan have shown high prevalence of A. baumannii as causative agent in cases of osteomyelitis secondary to traumatic injuries. Also, in Brazil, a retrospective study that analyzed 101 cases of osteomyelitis due to Gram-negative bacilli showed that A. baumannii was the second most prevalent agent, showing a high profile of antimicrobial resistance, particularly to carbapenems.

At the Institute of Orthopedics and Traumatology, Hospital das Clínicas, University of São Paulo, a Brazilian reference center that provides care for high-complexity orthopedic cases, 241 cases of osteomyelitis related to A. baumannii were treated between 2007 and 2014. All cases had microbiological confirmation, with positive cultures of bone tissue.

OBJECTIVES

1. Clinical and epidemiological characterization of 241 cases of osteomyelitis related to A. baumannii who were admitted at the Institute of Orthopedics and Traumatology, Hospital das Clínicas, University of São Paulo;
2. To describe the antimicrobial susceptibility profile of A. baumannii strains isolated;
3. To evaluate the patients' outcomes (remission, recurrence, limb amputation or death) according to the antimicrobial treatment used, including tigecycline.
4. To compare efficacy and safety profiles of tigecycline, colistin and ampicillin-sulbactan among patients with carbapenem-resistant A. baumannii related osteomyelitis.

METHODS This study will include data about all 241 patients with A. baumannii-related osteomyelitis admitted at our institution from 2007 to 2014. According to the institution´s protocol, diagnosis of osteomyelitis was based on the clinical history, infectious signs and symptoms and positive culture of bone tissue for A. baumannii. Bone samples were obtained from biopsy fragments identified as bone or medullary canal tissue (cortical bone and medullary canal aspirates) obtained through surgical procedures. All specimens were sent to the microbiology laboratory in thioglycolate culturing medium. The first reading was made 24 hours after incubation started and if the samples showed bacterial growth, the material was seeded in blood agar and MacConkey agar media. Bacterioscopic examinations were also performed. Subsequently, Gram-negative bacteria were identified by means of Vitek. Non-fermenting and Gram-positive bacteria were identified manually and a susceptibility test was performed using disk-diffusion. The minimum inhibitory concentrations were released in accordance with the CLSI criteria.

The following variables will be collected and analyzed for clinical characterization and outcomes evaluation:

* Gender;
* Age;
* Affected bones;
* Time of disease symptoms until hospital admission;
* Osteomyelitis-related symptoms;
* Previous antimicrobial use (before A. baumannii-positive culture);
* Classification of osteomyelitis (according to Waldwogel´s system);
* Presence of comorbidities (diabetes mellitus, active neoplasia, HIV infection, intravenous drug use, smoking, peripheral venous/arterial disease, alcoholism, open fracture, previous orthopedic surgery, imunossupressive conditions);
* ASA score;
* A. baumannii susceptibility profile;
* Antimicrobial drugs prescribed for A. baumannii-related infection;
* Antimicrobial drugs prescribed for concomitant infections;
* Antimicrobial-related side effects;
* Creatinine evolution following A. baumannii-related infection treatment;
* ESR, CPR and hemogram evolution following A. baumannii-related infection treatment;
* AST and ALT evolution following A. baumannii-related infection treatment;
* Radiological evolution of affected bone following A. baumannii-related infection treatment;
* Outcomes 6-month after A. baumannii-related infection treatment (disease remission, amputation of the affected limb, infection relapse, death and loss to follow-up). Disease remission will be defined as absence of signs of infection at the end of follow-up period.

Data analysis will be descriptive for all above mentioned variables among the 241 patients with A. baumanni-related osteomyelitis. Among those with infection related to carbapenem resistant-isolates, the variables concerning safety and efficacy of chosen antimicrobial regimen, colistin, ampicillin-sulbactan or tigeciclyne (antimicrobial-related side effects; creatinine evolution; ESR, CPR and hemogram evolution will be compared using chi-square test or Fisher's exact test for categoric variables and ANOVA test for continuous variables. Radiological variables and outcomes will be compared using chi-square test or Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

1. Microbiologically confirmed osteomyelitis related to Acinetobacter baumannii

Exclusion Criteria:

1. Impossibility to review data in medical records;
2. Culture results with A. baumannii considered as colonization.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include data about all 241 patients with A. baumannii-related osteomyelitis admitted at our institution from 2007 to 2014. According to the institution´s protocol, diagnosis of osteomyelitis was based on the clinical history, infectious signs and symptoms and bone tissue culturing that was positive for A. baumannii.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lucia L Lima, MD PhD, Principal Investigator — Associate Professor
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The initial database consisted of 262 patients. It was possible to collect data for 171 patients. Reasons for not including 91 patients:
  * non-location of medical records: 44;
  * culture results not considered for treatment: 29;
  * duplicate cases: 8;
  * other species of Acinetobacter: 7;
  * contamination / colonization: 3.
Groups:
- Carbapenem Susceptible A. Baumannii: 106 patients with osteomyelitis related to carbapenem-susceptible A. baumannii
- XDR Acinetobacter Baumannii: For this analysis, the 65 patients with XDR A. baumannii -related osteomyelitis, always resistant to carbapenems, treated with colistin or tigecycline were included.
Period: Overall Study
Arm/Group | Carbapenem Susceptible A. Baumannii | XDR Acinetobacter Baumannii
Started | 197 | 65
Completed | 106 | 65
Not Completed | 91 | 0
Not completed — non-location of medical records | 44 | 0
Not completed — culture results not considered for treat | 29 | 0
Not completed — duplicate cases | 8 | 0
Not completed — other species of Acinetobacte | 7 | 0
Not completed — contamination / colonization | 3 | 0

BASELINE CHARACTERISTICS:
Population: Patients with bone tissue culture positive for Acinetobacter baumannii submitted to surgical procedures to treat osteomyelitis.
Units Other Than Participants: Infections
Groups:
- Patients: All patients with bone tissue culture positive for Acinetobacter baumannii submitted to surgical procedures to treat osteomyelitis
Arm/Group | Patients
Number analyzed (Participants) | 171
Number analyzed (Infections) | 171
Age, Continuous [Mean (Full Range); unit: years] | 43.2 [6 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 134
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 171

OUTCOME MEASURES:

1. Primary Outcome: Description of the Clinical and Epidemiological Profile of Patients With Infection
Description: Distribution of the clinical and epidemiological characteristics studied among the patients. Use of percentage and average for description.
Time Frame: 6 months
Population: Described above.
Measure: Count of Participants; unit: Participants
Groups:
- Patients: Patients with A. baumannii-related osteomyelitis
Arm/Group | Patients
Number analyzed (Participants) | 171
Participants
  Remission | 92
  Relapse | 26
  Amputation | 25
  Lost follow-up | 21
  Death related to A. baumannii infection | 6
  Death not related to A. baumannii infection | 1

2. Secondary Outcome: A. Baumannii Susceptibility Profile
Description: A. baumannii isolates susceptible to the tested antimicrobials
Time Frame: 6 months
Population: Percentage of patients with carbapenem-susceptible isolates of A. baumannii
Measure: Count of Participants; unit: Participants
Groups:
- Susceptibility Profile of A. Baumannii Isolates Over Time: Variation in the susceptibility of A. baumannii isolates to antimicrobials over time from 2007 to 2015.
Arm/Group | Susceptibility Profile of A. Baumannii Isolates Over Time
Number analyzed (Participants) | 171
Participants | 57

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events (AE) reported within 48 hours after initiation of treatment with colistin (CL) or tigecycline (TG) were analysed: renal impairment;liver alterations; nausea/vomiting; and skin rash. Any other AE that occurred during treatment, was classified as "other event".
  AE were analyzed only for patients who received CL or TG. For this reason, there was no assessment of the occurrence of AE in patients in the "Carbapenem Susceptible A. baumannii" group, as they received neither CL nor TG.
Groups:
- XDR A. Baumannii: Patients with microbiologically proven XDR A. baumannii-related osteomyelitis who received colistin or tigecycline for treatment
Arm/Group | XDR A. Baumannii
All-Cause Mortality (participants affected / at risk) | 7/65
Serious Adverse Events (participants affected / at risk) | 36/65
Other Adverse Events (participants affected / at risk) | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XDR A. Baumannii (N=65)
Renal impairment (General disorders) | 27 (27) — Renal impairment
Liver abnormalities (Hepatobiliary disorders) | 2 (2) — Liver abnormalities
Nausea (Gastrointestinal disorders) | 4 (4) — Nausea
Skin rash (Immune system disorders) | 1 (1)
Other (Investigations) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03559530/Prot_SAP_000.pdf